CLINICAL TRIAL: NCT03804034
Title: Neurogenic Inflammation and Angiogenesis in the Human Dental Pulp in Response to Occlusal Interferences and Orthodontic Movements
Brief Title: Importance of Neurogenic Inflammation in the Angiogenic Response of the Dental Pulp as a Defensive Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institucion Universitaria Colegios de Colombia (Other)
Collaborators: Universidad Cooperativa de Colombia seccional Pasto (Unknown)
Responsible Party: Principal Investigator, Javier Caviedes-Bucheli, Endodontics postgraduate program professor, Cooperative University of Colombia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: JCB002
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Occlusal Trauma; Orthodontic Appliance Complication
Keywords: Neurogenic inflammation; Dental Pulp; Occlusal trauma; Orthodontics forces; SP; CGRP; VEGF
MeSH Terms: conditions — Neurogenic Inflammation

STUDY DESIGN:
Intervention Model Description: Human dental pulp was obtained from 40 freshly extracted maxillary and mandibular premolars with orthodontic indication from 20 healthy patients, both male and female, aged between 18 and 30 yearsThe premolars were randomly distributed into four groups, namely a group without occlusal trauma and orthodontic force chosen as the control group and three experimental groups, i.e., one occlusal trauma group experimentally induced by occlusal interferences, one moderate orthodontic force group, and one occlusal trauma plus moderate orthodontic force group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Occlusal trauma group (Experimental): an occlusal interference was placed on the lower teeth as follows. Articulating paper was used to mark the contact area between the upper and lower premolars indicated for extraction. Once established, the marked area on the lower premolar was acid-etched with 37% phosphoric acid for 15 s, washed, and dried. A bonding agent was placed and light-cured for 15 s, and finally, a 1- to 2-mm block of resin was placed over the contact area and light-cured for 40 s. Articulating paper was used again to verify that only the premolars that were going to be extracted had contact during normal occlusion as well as in lateral movements. Patients were given chewing gum and indications to repeat 20 masticatory cycles for 30 s, followed by a 30-s rest interval, and repeat the sequence again for a period of 30 min. This chewing cycle was repeated three times every 8 h for the first 24 h
  Interventions: Device: Block of resin
- Moderate orthodontic force group (Experimental): A convertible standard buccal tube was bonded over the buccal face of the first molar with resin and a McLaughlin, Bennett, and Trevisi slot size 0.022 bracket was bonded over the buccal face of the premolars. One 0.0017 × 0.025 in titanium molybdenum alloy wire cantilever was inserted into each first molar tube, and the wire was bent buccally to form a helix. The cantilever was clinched to the distal end of the tube, and a tipping and extrusive force was applied on the premolar. The activation angle was 45° with a force of 56 g, which was applied to the tooth for 24 h before it was extracted.
  Interventions: Device: Buccal tube, Bracket and 0.0017 × 0.025 in titanium molybdenum alloy wire
- Occlusal trauma and moderate orthodontic force group (Experimental): the combination of occlusal trauma and orthodontic force .
  Interventions: Device: Block of resin; Device: Buccal tube, Bracket and 0.0017 × 0.025 in titanium molybdenum alloy wire
- Control Group (No Intervention): No experimental device to produce occlusal trauma or orthodontic forces

INTERVENTIONS:
Device: Block of resin
  Arms: Occlusal trauma and moderate orthodontic force group; Occlusal trauma group
Device: Buccal tube, Bracket and 0.0017 × 0.025 in titanium molybdenum alloy wire
  Arms: Moderate orthodontic force group; Occlusal trauma and moderate orthodontic force group

SUMMARY:
This study measures SP, CGRP and VEGF expression in human dental pulp under occlusal trauma induced by occlusal interferences under moderate orthodontic forces or under a combination of occlusal trauma and moderate orthodontic forces because in clinical reality, patients under orthodontic treatment experience a combination of these stimuli on their pulp tissue.

DETAILED DESCRIPTION:
Substance P (SP) and calcitonin gene-related peptide (CGRP) are neuropeptides that are assembled in the cell bodies of the trigeminal nerve and are transported through axonal flow to the nerve endings in human dental pulp, mainly in type-C nerve fibers and free nerve endings, where they are released to fulfill important biological functions.

SP plays an important role in pulp tissue reparation because it stimulates angiogenesis using direct mechanisms by modulating the growth of endothelial cells and fibroblasts through the activation of growth factors such as VEGF and IGF-1 and stimulates cell migration and proliferation to form mineralized tissue as a defense mechanism. It also uses indirect mechanisms such as binding to granulocytes or macrophages, which allow cells with angiogenic potential to be attracted.

CGRP has a key role in pulp reparation because of its angiogenic potential, which is linked to endothelial cell stimulation via the cAMP-PKA pathway, promoting cell proliferation. It boosts VEGF expression and stimulates focal adhesion kinase involved in the stabilization and maturation of blood vessels. It can stimulate growth factors that act on fibroblasts, such as HGF, IGF-1, and bFGF, and it can also produce an effect on odontoblast-like cells by increasing BMP-2 expression and allowing cell proliferation after 24 h. This shows that it can contribute to mineralized matrix formation

Angiogenesis is mediated by several growth factors, such as the VEGF. VEGF is released in the pulp tissue as a response to a harmful stimulus to counteract emerging hypoxic areas regulating oxygen and nutrients supply to cell populations by forming new blood vessels. VEGF is present in endothelial cells, mast cells, macrophages, lymphocytes, undifferentiated mesenchymal cells, fibroblasts, and odontoblast-like cells, and it controls neurogenic inflammation and reparation processes in combination with SP due to its angiogenic potential.

SP, CGRP, VEGF expression can be altered by the masticatory function, occlusal trauma, orthodontic movements, or a combination of occlusal trauma and orthodontic movements, which often takes place in patients under orthodontic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Teeth in normal masticatory function
* Complete root development verified clinically and radiographically

Exclusion Criteria:

* Patients under medication
* Smokers
* Pregnant women were excluded
* Teeth with caries
* Teeth with restaurations,
* Teeth with previous orthodontic treatment
* Teeth with periodontal disorders
* Teeth with parafunctional habits.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-07-02 (Actual); Primary Completion 2014-01-27 (Actual); Study Completion 2015-01-12 (Actual)

PRIMARY OUTCOMES:
SP expression (pmol/mg in pulp tissue) | 24 hours stimulations
  Sample Collection: All the teeth involved in this study were anesthetized and extracted 5 min after anesthetic application with conventional methods. Immediately after extraction, teeth were sectioned. Pulp tissue was obtained using a sterile endodontic excavator, placed on an Eppendorf tube, snap frozen in liquid nitrogen until the radioimmunoassay (RIA) test was performed.
  Results are presented as SP expression in pmol/mg of pulp tissue. Means and standard deviations as well as minimum and maximum values for each neuropeptide were calculated.

SECONDARY OUTCOMES:
CGRP expression (pmol/mg in pulp tissue) | 24 hours stimulations
  Sample Collection: All the teeth involved in this study were anesthetized and extracted 5 min after anesthetic application with conventional methods. Immediately after extraction, teeth were sectioned. Pulp tissue was obtained using a sterile endodontic excavator, placed on an Eppendorf tube, snap frozen in liquid nitrogen until the radioimmunoassay (RIA) test was performed.
  Results are presented as CGRP expression in pmol/mg of pulp tissue. Means and standard deviations as well as minimum and maximum values for each neuropeptide were calculated.
VEGF expression (pmol/mg in pulp tissue) | 24 hours stimulations
  Sample Collection: All the teeth involved in this study were anesthetized and extracted 5 min after anesthetic application with conventional methods. Immediately after extraction, teeth were sectioned. Pulp tissue was obtained using a sterile endodontic excavator, placed on an Eppendorf tube, snap frozen in liquid nitrogen until the radioimmunoassay (RIA) test was performed.
  Results are presented as CGRP expression in pmol/mg of pulp tissue. Means and standard deviations as well as minimum and maximum values for each growth factor were calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Odontologia, Unicoc, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benemei S, Nicoletti P, Capone JG, Geppetti P. CGRP receptors in the control of pain and inflammation. Curr Opin Pharmacol. 2009 Feb;9(1):9-14. doi: 10.1016/j.coph.2008.12.007. Epub 2009 Jan 20. PMID 19157980
- [Background] Caviedes-Bucheli J, Arenas N, Guiza O, Moncada NA, Moreno GC, Diaz E, Munoz HR. Calcitonin gene-related peptide receptor expression in healthy and inflamed human pulp tissue. Int Endod J. 2005 Oct;38(10):712-7. doi: 10.1111/j.1365-2591.2005.01006.x. PMID 16164685
- [Background] Caviedes-Bucheli J, Azuero-Holguin MM, Correa-Ortiz JA, Aguilar-Mora MV, Pedroza-Flores JD, Ulate E, Lombana N, Munoz HR. Effect of experimentally induced occlusal trauma on substance p expression in human dental pulp and periodontal ligament. J Endod. 2011 May;37(5):627-30. doi: 10.1016/j.joen.2011.02.013. PMID 21496661
- [Background] Caviedes-Bucheli J, Gomez-Sosa JF, Azuero-Holguin MM, Ormeno-Gomez M, Pinto-Pascual V, Munoz HR. Angiogenic mechanisms of human dental pulp and their relationship with substance P expression in response to occlusal trauma. Int Endod J. 2017 Apr;50(4):339-351. doi: 10.1111/iej.12627. Epub 2016 Apr 2. PMID 26953220
- [Background] Caviedes-Bucheli J, Lombana N, Azuero-Holguin MM, Munoz HR. Quantification of neuropeptides (calcitonin gene-related peptide, substance P, neurokinin A, neuropeptide Y and vasoactive intestinal polypeptide) expressed in healthy and inflamed human dental pulp. Int Endod J. 2006 May;39(5):394-400. doi: 10.1111/j.1365-2591.2006.01093.x. PMID 16640639
- [Background] Saghiri MA, Asatourian A, Sorenson CM, Sheibani N. Role of angiogenesis in endodontics: contributions of stem cells and proangiogenic and antiangiogenic factors to dental pulp regeneration. J Endod. 2015 Jun;41(6):797-803. doi: 10.1016/j.joen.2014.12.019. Epub 2015 Jan 31. PMID 25649306
- [Background] Wei F, Yang S, Xu H, Guo Q, Li Q, Hu L, Liu D, Wang C. Expression and Function of Hypoxia Inducible Factor-1alpha and Vascular Endothelial Growth Factor in Pulp Tissue of Teeth under Orthodontic Movement. Mediators Inflamm. 2015;2015:215761. doi: 10.1155/2015/215761. Epub 2015 Sep 9. PMID 26441483
- [Background] Potente M, Gerhardt H, Carmeliet P. Basic and therapeutic aspects of angiogenesis. Cell. 2011 Sep 16;146(6):873-87. doi: 10.1016/j.cell.2011.08.039. PMID 21925313
- [Result] Awawdeh L, Lundy FT, Shaw C, Lamey PJ, Linden GJ, Kennedy JG. Quantitative analysis of substance P, neurokinin A and calcitonin gene-related peptide in pulp tissue from painful and healthy human teeth. Int Endod J. 2002 Jan;35(1):30-6. doi: 10.1046/j.1365-2591.2002.00451.x. PMID 11853236
- [Derived] Caviedes-Bucheli J, Lopez-Moncayo LF, Munoz-Alvear HD, Gomez-Sosa JF, Diaz-Barrera LE, Curtidor H, Munoz HR. Expression of substance P, calcitonin gene-related peptide and vascular endothelial growth factor in human dental pulp under different clinical stimuli. BMC Oral Health. 2021 Mar 23;21(1):152. doi: 10.1186/s12903-021-01519-x. PMID 33757513